CLINICAL TRIAL: NCT03976180
Title: A Multicentre, Prospective, Randomized, Multi-arm, Multi-stage Clinical Trial of High-flow Oxygen for Vaso-occlusive Pain Crisis in Adult Patients With Sickle Cell Disease;
Brief Title: High-flow Oxygen for Vaso-occlusive Pain Crisis
Acronym: OSONE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fisher and Paykel Healthcare (Industry); Orkyn' (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P180303J
Record Dates: First submitted 2019-05-24; First posted 2019-06-05 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2024-10

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; vaso-occlusive pain crisis; HFNO; ACS
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This is a comparative randomized controlled superiority open-label multi-arm multi-stage (MAMS) trial. The study will use a multi-arm multi-stage (MAMS) trial design with three stages and four arms (one control arm and three intervention arms).
  * "Pilot" stage: a formal safety/feasibility testing. Research arms will only continue to recruitment in the next stage if they have been shown to be both safe and feasible, although patient data from all patients and all stages will be included in the final analyses.
  * "Activity" stage: an interim comparison of activity using the rate of VOC resolution without complication at day-5 as primary endpoint. At the end of this stage, an interim analysis will be used in order to select the most promising experimental treatment and compare it to control in the subsequent stage ("pick the winner" strategy).
  * "Efficacy" stage: final comparison with secondary ACS at day-14 as the primary endpoint.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- standard low-flow oxygen (Active Comparator): In the control group, standard low-flow oxygen will be delivered via nasal prongs (LFNO), up to hospital discharge or secondary ACS onset, in order to achieve normoxia (target pulse oxymetry saturation of 95%). This strategy is in accordance with current recommendations and usual care;
  Interventions: Device: Stadard low-flow oxygen
- HFNO with low FiO2 (21%-30%) (Experimental): HFNO with low FiO2 (21%-30%) targeting normoxia: to test the effect of improved pulmonary function;
  Interventions: Device: HFNO with low FiO2 (21%-30%)
- HFNO with intermediate FiO2 (50%) (Experimental): HFNO with intermediate FiO2 (50%): to test the combined effect of improved pulmonary function and moderate hyperoxia; in this group, FiO2 will be set at 50% during the first 24 hours of intervention to target moderate hyperoxia, then reduced to 21-30% during the following 48 hours to target normoxia
  Interventions: Device: HFNO with intermediate FiO2 (50%)
- HFNO with high FiO2 (100%) (Experimental): HFNO with high FiO2 (100%): to test the combined effect of improved pulmonary function and intense hyperoxia; in this group, FiO2 will be set at 100% during the first 24 hours of intervention to target intense hyperoxia, then reduced to 21-30% during the following 48 hours to target normoxia
  Interventions: Device: HFNO with high FiO2 (100%)

INTERVENTIONS:
Device: Stadard low-flow oxygen — In the control group, standard low-flow oxygen will be delivered via nasal prongs (LFNO), up to hospital discharge or secondary ACS onset, in order to achieve normoxia (target pulse oxymetry saturation of 95%). This strategy is in accordance with current recommendations and usual care
  Other Names: Control group
  Arms: standard low-flow oxygen
Device: HFNO with low FiO2 (21%-30%) — HFNO with low FiO2 (21%-30%) targeting normoxia: to test the effect of improved pulmonary function
  Other Names: Intervention group
  Arms: HFNO with low FiO2 (21%-30%)
Device: HFNO with intermediate FiO2 (50%) — In this group, FiO2 will be set at 50% during the first 24 hours of intervention to target moderate hyperoxia, then reduced to 21-3025% during the following 48 hours to target normoxia
  Other Names: Intervention group
  Arms: HFNO with intermediate FiO2 (50%)
Device: HFNO with high FiO2 (100%) — In this group, FiO2 will be set at 100% during the first 24 hours of intervention to target intense hyperoxia, then reduced to 21-3025% during the following 48 hours to target normoxia
  Other Names: Intervention group
  Arms: HFNO with high FiO2 (100%)

SUMMARY:
Sickle cell disease (SCD) is characterized by recurrent vaso-occlusive pain crisis (VOC), which may evolve to acute chest syndrome (ACS), the most common cause of death among adult patients with SCD. Currently, there is no safe and effective treatment to abort VOC or prevent secondary ACS. Management of VOC mostly involve a symptomatic approach including hydration, analgesics, transfusion, and incentive spirometry, which was investigated in a very limited number of patients (<30).

The polymerisation of HbS is one major feature in the pathogenesis of vaso-occlusion. Among factors determining the rate and extent of HbS polymer formation, the hypoxic stimulus is one of the most potent and readily alterable. Current guidelines recommend oxygen therapy in patients with VOC in order to maintain a target oxygen saturation of 95%. Low-flow nasal oxygen (LFNO) is routinely used to achieve this normoxia approach, particularly in patients at risk of secondary ACS because they may experience acute desaturation. In contrast, various case series suggest a potential beneficial role of intensified oxygen therapy targeting hyperoxia for the management of VOC, particularly with the use of hyperbaric oxygen, but the latter is difficult to implement in routine clinical practice.

A recent high-flow nasal oxygen (HFNO) technology allows the delivery of humidified gas at high fraction of inspired oxygen (FiO2) through nasal cannula. The FiO2 can be adjusted up to 100% (allowing hyperoxia that may reverse sickling) and the flow can be increased up to 60 L/min (which generates positive airway pressure and dead space flushing, that may prevent evolution of VOC towards ACS by alleviating atelectasis and opioid-induced hypercapnia). In patients with acute respiratory failure, HFNO has been shown to improve patient's comfort, oxygenation, and survival as compared to standard oxygen or non-invasive ventilation.

The aim of the present study is to test the efficacy and safety of HFNO for the management of VOC and prevention of secondary ACS. The investigators will use a multi-arm multi-stage (MAMS) design to achieve these goals. HFNO will be delivered through AIRVO 2 (Fisher and Paykel Healthcare, New Zealand), a device that incorporates a turbine allowing its use in hospital wards.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Patient with major sickle cell disease syndrome (SS, SC, Sβ0 or Sβ+);
* VOC as defined by acute pain or tenderness, affecting at least one part of the body, including limbs, ribs, sternum, head (skull), spine, and/or pelvis, that requires opioids and is not attributable to other causes;
* Intermediate-to-high risk for secondary ACS derived from the PRESEV score (Bartolucci et al, EBioMedicine 2016) as follows: a reticulocyte count >216 G/L OR at least two of the followings : i) spine and/or pelvis CPS >1; ii) leucocyte count >11G/L; iii) hemoglobin ≤ 9 g/dL; in case of long-term treatment by hydroxyurea, only one of the above mentioned criteria will be needed, given its effects on hemoglobin, leucocyte and reticulocytes counts;
* Informed consent;
* Patient affiliated to social security

Exclusion Criteria:

The presence at inclusion of a primary ACS. Primary ACS is defined by the combination at time of randomization of a clinical sign [chest pain or auscultatory abnormality (crepitants and/or bronchial breathing)] with a new pulmonary infiltrate (on chest film, thoracic scan, or lung ultrasound);

* VOC with need of parenteral opioids lasting longer than 72 hours at time of inclusion;
* Known pregnancy or current lactation; Women of child bearing potential will be tested for pregnancy before inclusion;
* Known cerebral vasculopathy or past medical history of stroke, due to Moya Moya or persisting visible macrovessel stenosis/occlusion;
* Known ischemic heart disease or typical chest angina;
* Patient who is currently enrolled in other investigational drug study;
* Known legal incapacity,
* Prisoners or subjects who are involuntarily incarcerated
* Anatomical factors precluding placement of a nasal cannula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2020-04-27 (Actual); Primary Completion 2025-11-27 (Estimated); Study Completion 2025-11-27 (Estimated)

PRIMARY OUTCOMES:
Rate of cardiac and neurologic related events (Pilot Stage) | At the end end of the "pilot stage" and up to 28 days
  This endpoint will be assessed at the end of the "pilot stage" and throughout the entire study for cumulative safety information. Research arms will only continue to recruitment in the next stage if they have been shown to be both safe (<5 cardiac or neurologic related events, in the arm during the pilot phase as defined by one of the following: acute coronary syndrome, acute ischemic stroke, or seizure) and feasible (<8 definitive discontinuations before day-2 due to patient's intolerance), although patient data from all patients and all stages will be included in the final analyses.
Rate of vaso-occlusive pain crisis (VOC) resolution without complication (Activity stage) | Day 5
  VOC will be considered terminated when at least 3 of the following 4 criteria are met at two consecutive assessments: i) absence of fever for 8 hours; ii) absence of pain progression and no requirement of intravenous infusion of opioid analgesics for the last 8 hours; iii) the patient is able to walk or move without pain; iv) absence of spontaneous pain with a CPS (categorical pain score) of 1 or less
Rate of secondary acute chest syndrome (ACS)(Efficacy Stage) | Day 14
  Defined as the proportion of patients with secondary ACS during the 14 days following randomization. Secondary ACS is defined as the combination after randomization of a clinical sign [chest pain or auscultatory abnormality (crepitants and/or bronchial breathing)] with a new pulmonary infiltrate (on chest film, thoracic scan, or lung ultrasound).

SECONDARY OUTCOMES:
Volume of transfused red blood cells and volume of exsanguinated blood | Between day-1 (randomization) and day-14
Pain intensity evaluated by categorical pain score | Between day-1 (randomization) and day-14
  Pain intensity evaluated with categorical pain score (CPS). Patients will grade their pain (range 0-3 points, with 0, no pain; 1, mild pain, unaffected by mobilization; 2, moderate pain, increased by mobilization; 3, severe pain with disability) in seven body sites (all four limbs, ribs and sternum, head, and spine and pelvis)
Pain intensity evaluated by visual analogue scale | Between day-1 (randomization) and day-14
  Pain intensity evaluated with the visual analogue pain scale (VAS) .It is presented as a 10 cm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "no pain at all" and "worst pain imaginable."
VOC duration | Day-14
VOC-free days | Day-14
Reticulocyte count | Day-2 and Day-5
Arterial blood gas | Up to 24 hours
  Arterial blood gas assessed at least once during the first 24 hours of treatment (if available)
Cumulative doses of intravenous and subcutaneous opioids | Between day-1 (randomization) and day-14
Number of complicated VOC | Day-14
  A complicated VOC is defined as the occurrence of at least one of the following events between randomization and day-14: transfusion, exchange transfusion, mechanical ventilation, shock (catecholamine infusion), intensive care admission or death.
Duration of hospital stay | Day-28
  Defined as the time from randomization to hospital discharge; patients still hospitalized at day-28 will be attributed a hospital stay of 28 days)
Number of re-hospitalizations or emergency department consultations for VOC or ACS | Up to 28 days
Number of death (Mortality) | Day-28

CONTACTS AND LOCATIONS:
Overall Officials: Armand Mekontso, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor, Créteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION

REFERENCES:
- [Derived] Mekontso Dessap A, Habibi A, Guillaud C, Kassasseya C, Larrat C, Agbakou M, Tchoubou T, Candille C, Carpentier B, Landais M, Arlet JB, Fartoukh M, Desclaux A, Masseau A, Oziel J, Bouharaoua S, Affo C, Viglino D, Boukari L, Martin LE, Ngo S, Anguel N, Chantalat C, Bourgarit-Durand A, Genty I, Makowski C, Guillet S, Melica G, Lionnet F, Le Jeune S, Joseph L, Lanternier F, Cougoul P, Bertchansky I, Boue Y, Bartolucci P, Gendreau S, Audureau E. High flow oxygen for vaso-occlusive crisis: a multicentre, prospective, randomised, multi-arm, multi-stage clinical trial (OSONE). BMJ Open. 2025 Sep 17;15(9):e104564. doi: 10.1136/bmjopen-2025-104564. PMID 40967654